CLINICAL TRIAL: NCT00815646
Title: Effects of the Dive Reflex on Pulmonary Arterial and Pulmonary Artery Wedge Pressures in Subjects Who Have Experienced Immersion Pulmonary Edema
Brief Title: Prevention and Treatment of Immersion Pulmonary Edema
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Divers Alert Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00003158
Record Dates: First submitted 2008-12-26; First posted 2008-12-30 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Immersion Pulmonary Edema (IPE); Swimming Induced Pulmonary Edema (SIPE)
Keywords: Immersion pulmonary edema; Diving; Swimming; Pulmonary edema; Cold water immersion
MeSH Terms: conditions — Pulmonary Edema | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil (Experimental): Measurements of pulmonary and systemic pressures during cold water immersion before and after sildenafil 50 mg orally.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — After measurement of the effect of cold water on cardiac output and pulmonary artery and wedge pressures, a single dose of sildenafil (50 mg) will be given orally, followed by similar hemodynamic measurements.
  Other Names: Viagra

SUMMARY:
Immersion pulmonary edema (IPE) is a condition in which fluid fills the lungs during diving or swimming, particularly in cold water. Some individuals appear to be predisposed to developing IPE. DNA samples will be collected and stored, in order to compare the genetic profiles of individuals who have experienced IPE with those who have not. In a few individuals who have experienced IPE, we plan to measure the effects of cold water immersion on the blood pressure, cardiac output and the pressures in the pulmonary artery. These will be compared with similar measurements already obtained from normal individuals.

DETAILED DESCRIPTION:
Immersion pulmonary edema (IPE) is a condition that has sudden onset in swimmers and divers, and is characterized by cough, shortness of breath, decreased blood oxygen levels, and hemoptysis. The purpose of this study is to examine the effects of cold water immersion and the dive reflex on pulmonary arterial pressure and pulmonary capillary wedge pressure in those who have already experienced IPE, as well as explore the possibility of a genetic predisposition. Healthy nonsmoking subjects who have experienced IPE will be recruited for several cold-water immersion experiments and DNA analysis. Their pulmonary arterial and pulmonary arterial wedge pressures will be measured as they undergo immersed rest and exercise trials in thermoneutral and cold water. If the pressures increase with these trials as hypothesized, the effects of sildenafil administration (a pulmonary vasodilator) will be tested during a second trial. Blood will also be drawn for DNA analysis of certain genes with possible relation to IPE. Results of these tests will be compared with those of the general population.

ELIGIBILITY:
Inclusion Criteria:

* History of immersion pulmonary edema

Exclusion Criteria:

* Coronary artery disease, cardiomyopathy, heart valve disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery pressure during cold water immersion | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Peacher DF, Pecorella SR, Freiberger JJ, Natoli MJ, Schinazi EA, Doar PO, Boso AE, Walker AJ, Gill M, Kernagis D, Uguccioni D, Moon RE. Effects of hyperoxia on ventilation and pulmonary hemodynamics during immersed prone exercise at 4.7 ATA: possible implications for immersion pulmonary edema. J Appl Physiol (1985). 2010 Jul;109(1):68-78. doi: 10.1152/japplphysiol.01431.2009. Epub 2010 Apr 29. PMID 20431020
- [Background] Fraser JA, Peacher DF, Freiberger JJ, Natoli MJ, Schinazi EA, Beck IV, Walker JR, Doar PO, Boso AE, Walker AJ, Kernagis DN, Moon RE. Risk factors for immersion pulmonary edema: hyperoxia does not attenuate pulmonary hypertension associated with cold water-immersed prone exercise at 4.7 ATA. J Appl Physiol (1985). 2011 Mar;110(3):610-8. doi: 10.1152/japplphysiol.01088.2010. Epub 2010 Dec 9. PMID 21148341
- [Background] Peacher DF, Martina SD, Otteni CE, Wester TE, Potter JF, Moon RE. Immersion pulmonary edema and comorbidities: case series and updated review. Med Sci Sports Exerc. 2015 Jun;47(6):1128-34. doi: 10.1249/MSS.0000000000000524. PMID 25222821
- [Derived] Moon RE, Martina SD, Peacher DF, Potter JF, Wester TE, Cherry AD, Natoli MJ, Otteni CE, Kernagis DN, White WD, Freiberger JJ. Swimming-Induced Pulmonary Edema: Pathophysiology and Risk Reduction With Sildenafil. Circulation. 2016 Mar 8;133(10):988-96. doi: 10.1161/CIRCULATIONAHA.115.019464. Epub 2016 Feb 16. PMID 26882910
- See also: Duke Center for Hyperbaric Medicine and Environmental Physiology — http://dukedivemedicine.org/?p=1656